CLINICAL TRIAL: NCT02434822
Title: Safety and Immunogenicity of Two Doses of Oral Cholera Vaccine (ShancholTM) in Subjects Aged 1 Year and Older in Dominican Republic
Brief Title: A Study of Two Doses of Oral Cholera Vaccine (Shanchol™) in Subjects Aged 1 Year and Older in Dominican Republic
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SHC03; U1111-1127-7355 (Other: WHO)
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Cholera
Keywords: Cholera; Shanchol™; Cholera Vaccine
MeSH Terms: conditions — Cholera | interventions — shanchol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Study Group 1 (Experimental): Participants aged 1 through 4 years at enrollment
  Interventions: Biological: Shanchol™: Oral Cholera Vaccine Killed Bivalent (O1 and O139) Whole Cell
- Study Group 2 (Experimental): Participants aged 5 through 14 years at enrollment
  Interventions: Biological: Shanchol™: Oral Cholera Vaccine Killed Bivalent (O1 and O139) Whole Cell
- Study Group 3 (Experimental): Participants aged 15 years and above at enrollment
  Interventions: Biological: Shanchol™: Oral Cholera Vaccine Killed Bivalent (O1 and O139) Whole Cell

INTERVENTIONS:
Biological: Shanchol™: Oral Cholera Vaccine Killed Bivalent (O1 and O139) Whole Cell — 1.5 mL, Oral administration
  Other Names: Shanchol™
  Arms: Study Group 1
Biological: Shanchol™: Oral Cholera Vaccine Killed Bivalent (O1 and O139) Whole Cell — 1.5 mL, Oral administration
  Other Names: Shanchol™
  Arms: Study Group 2
Biological: Shanchol™: Oral Cholera Vaccine Killed Bivalent (O1 and O139) Whole Cell — 1.5 mL, Oral administration
  Other Names: Shanchol™
  Arms: Study Group 3

SUMMARY:
The aim of the study is to generate safety and immunogenicity data with Shanchol in The Philippines

Objectives:

* To describe the safety after each dose of Shanchol vaccine.
* To describe the immunogenicity after each dose of Shanchol vaccine.

DETAILED DESCRIPTION:
Healthy study participants aged 1 year and older will receive two doses of vaccine 14 days apart, and will be assessed baseline immunogenicity (pre-vaccination) and 14 days after each vaccine dose. Safety data will be collected for 14 days after the first dose and 30 days after the second dose.

ELIGIBILITY:
Inclusion Criteria:

* Aged 1 year and older on the day of inclusion
* Subjects aged 1 through 17 years: Informed consent form has been signed and dated by the parent(s) or another legally acceptable representative and assent form has been signed and dated by the subject if aged 9 through 17 years Subjects aged 18 years and older: Informed consent form has been signed and dated by the subject
* Subjects and/or subject's parent or an adult family member delegated by parent / legally acceptable representative are able to attend all scheduled visits and to comply with all trial procedures
* Subjects aged less than 2 years only: Born at full term of pregnancy (≥ 37 weeks) and/or with a birth weight ≥ 2.5 kg.

Exclusion Criteria:

* Subject is pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be pre-menarche or post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination and until at least 4 weeks after the last vaccination)
* Participation at the time of study enrollment or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination or planned receipt of any vaccine in the 4 weeks following any trial vaccination except for influenza vaccination, which may be received at least 2 weeks before or after any study vaccination
* Previous vaccination against cholera (in the previous 5 years) with either the trial vaccine or another vaccine
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* History of cholera infection, confirmed either clinically, serologically, or microbiologically
* At high risk for cholera infection during the trial (i.e., subject residing in areas with poor sanitary conditions)
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Intake of oral antibiotics within one week prior to enrollment
* Moderate or severe acute illness / infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 38.0°C). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* Identified as an Investigator or employee of the Investigator / study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study
* Diarrhea (3 or more loose/watery stools within a 24-hours period) within 6 weeks prior to enrollment. A prospective subject should not be included in the study until the condition has resolved
* Intake of anti-diarrhea medicine within one week prior to enrollment
* Abdominal pain or cramps, loss of appetite, nausea, or vomiting within 24 hours prior to enrollment. A prospective subject should not be included in the study until the condition has resolved.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of participants reporting unsolicited systemic adverse events (AEs); solicited systemic reactions including serious adverse events following administration Oral Cholera Vaccine (Shanchol™) | Day 0 up to Day 44 post oral vaccination
  Solicited systemic reaction: Vomiting, Diarrhea, Fever (temperature), Abdominal pain, Itching, Rash, Weakness, Cough, Vertigo, and Dryness of Mouth
Summary of titers of serum vibriocidal antibodies Before and 14 days after each Oral Cholera Vaccine (Shanchol™) | Day 0 (before) and Day 14 Post oral vaccination
  Serum vibriocidal antibody (against V. cholerae O1 Inaba serogroup, V. cholerae O1 Ogawa serogroup, and V. cholerae O139 serogroup) will be assessed using the microtiter technique.

SECONDARY OUTCOMES:
Number of participants with 4-fold or greater rises in titers 14 days after each Oral Cholera Vaccine (Shanchol™) relative to baseline | Day 0 (before) and Day 14 Post oral vaccination
  Serum vibriocidal antibody (against V. cholerae O1 Inaba serogroup, V. cholerae O1 Ogawa serogroup, and V. cholerae O139 serogroup) will be assessed using the microtiter technique.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (1):
- Santo Domingo, Dominican Republic

REFERENCES:
- [Result] Cordero De Los Santos L, Feris-Iglesias J, Aloysia D'Cor N, Midde VJ, Patnaik BN, Thollot Y, Rasuli A, Desauziers E. Bivalent oral cholera vaccine in participants aged 1 year and older in the Dominican Republic: A phase III, single-arm, safety and immunogenicity trial. Hum Vaccin Immunother. 2018 Jun 3;14(6):1403-1411. doi: 10.1080/21645515.2018.1430540. Epub 2018 Feb 22. PMID 29470934